CLINICAL TRIAL: NCT02753257
Title: Validation of Sensitivity and Specificity of a Multi-Omic Precision Diagnostic for Acute Stroke Evaluation (VALISS)
Brief Title: Validation of Sensitivity and Specificity of a Multi-Omic Precision Diagnostic for Acute Stroke Evaluation
Acronym: VALISS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Valtari Bio (Industry)
Collaborators: University of Cincinnati (Other); University of Texas at Austin (Other)
Responsible Party: Sponsor
Other Study IDs: ValtariBio-5-01
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Stroke
Keywords: stroke; stroke mimic
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples will be collected from all patients at baseline resulting in two 2.5 ml Paxgene RNA tubes, two 8 ml EDTA tube, and one 7 ml serum tube. Approximately 28 ml of blood will be collected.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
Valtari Bio has early proof of concept clinical data of a multi-omic peripheral blood biomarker profile that can be used to determine stroke from no stroke in the emergency setting. The objective of this observational cohort clinical study is to determine the clinical utility of this multi-omic biomarker profile.

Primary Study Aims:

1. The diagnostic tests characteristics of a multi-omic biomarker diagnostic for stroke (ischemic stroke, transient ischemic attack (TIA) and hemorrhagic stroke) versus no stroke (stroke mimic).
2. The ability of a multi-omic biomarker profile to differentiate ischemic stroke from hemorrhagic stroke and TIA.

DETAILED DESCRIPTION:
At the completion of this project the investigators will have evaluated a peripheral blood test that determines the expression of a multi-omic biomarker profile to differentiate stroke from no-stroke in the emergency setting. Five hundred patients aged 18 years or older who present to the hospital with stroke-like symptoms will be recruited within 24 hours of symptom onset at participating clinical sites. Data will be obtained from the medical records. Blood for research purposes will be obtained. Research evaluations for stroke severity, symptoms and outcome will be performed by trained personnel. All clinical evaluation and management will be per standard of care.

The primary outcome of this study is the criterion standard stroke diagnosis. This will be used to estimate the diagnostic test characteristics of a multi-omic biomarker profile in the peripheral whole blood for distinguishing stroke (IS, TIA, SAH, ICH) versus non-stroke in ED patients with acute neurologic symptoms. Secondly, the investigators will estimate the ability of the multi-omic biomarker profile to differentiate between stroke subtypes. A diagnosis of stroke will be defined as clinical syndromes consistent with stroke (i.e., sudden onset neurological deficit) plus imaging confirmation (or symptom resolution and lack of imaging findings in TIA). Finally, the investigators will explore the relationship between the multi-omic profile and time from symptom onset in ischemic stroke patients. Descriptive and inferential statistics will be used to address the aims of the study. Pattern recognition analysis and machine learning will be employed as a systems level approach to determine relevant pathophysiologic pathways associated with diagnosis and symptom onset time.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older who present with symptoms of a possible stroke in whom blood can be collected for this study within 12 hours of symptom onset will be eligible.

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective consecutive sample of possible stroke cases will be recruited within 12 hours of symptom onset. Final diagnoses may include: ischemic stroke (IS), TIA, aneurysmal subarachnoid hemorrhage (SAH), intracerebral hemorrhage (ICH) with or without intraventricular hemorrhage (IVH) (or primary IVH), and stroke mimic (all other patients presenting with acute onset stroke-like symptoms who do not have ischemic or hemorrhagic stroke).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically definite ischemic stroke (focal neurological deficits persisting for more than 24 hours) confirmed by non-investigational CT or MRI | within the first 24 hours of emergency evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Taura L Barr, PhD RN, Principal Investigator — Valtari Bio
Locations (2):
- United States (2):
  - University of Cincinnati University Hospital, Cincinnati, Ohio
  - University of Texas at Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes